CLINICAL TRIAL: NCT03850600
Title: The MELODY Trial: Modulating Early Life Microbiome Through Dietary Intervention in Crohn's Disease
Brief Title: Modulating Early Life Microbiome Through Dietary Intervention in Crohn's Disease
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: The Leona M. and Harry B. Helmsley Charitable Trust (Other); University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Inga Peter, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GCO 18-2246
Record Dates: First submitted 2019-02-15; First posted 2019-02-22 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2024-11

CONDITIONS: Crohn Disease; Pregnancy
Keywords: Microbiota; Diet; Immune System
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Intervention Model Description: The study design is a three-arm, prospective, pre-post intervention trial. Crohn's Disease (CD) patients at 27-29 weeks of pregnancy will self-select to Arm 1 or Arm 2. Controls will be in Arm 3.
  1. Arm 1 (diet-CD): 8-10 weeks of dietary intervention (n=66)
  2. Arm 2 (no-diet-CD): usual diet with no intervention (n=66)
  3. Arm 3 (no-diet-control): unaffected controls at the same gestational stage will follow their usual diet and no intervention (n=66).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Diet-CD (Experimental): dietary intervention: 8-10 weeks of diet intervention
  Interventions: Other: Diet-CD
- No-Diet-CD (No Intervention): Usual diet with no intervention
- No-Diet-Control (No Intervention): Unaffected controls at the same gestational stage will follow usual diet and no intervention

INTERVENTIONS:
Other: Diet-CD — CD patients will self-select into the intervention arm to follow the diet for 8-10 weeks during their third trimester of pregnancy.
  Other Names: Diet Arm
  Arms: Diet-CD

SUMMARY:
The MELODY Trial: Modulating Early Life Microbiome through Dietary Intervention in Crohn's Disease, will test whether a non-invasive dietary intervention during pregnancy can improve the gut microbiota composition in both pregnant Crohn's disease patients and their babies during the sensitive time window of infant immune system development, and whether this can lead to decreased risk of maternal disease relapse postpartum and decreased functional gastrointestinal disorders and gut inflammation in their babies. Through this trial, the study team hopes to better understand the origin of the initial gut bacterial colonization in babies, providing potential intervention targets to prevent Crohn's disease development in high risk individuals.

DETAILED DESCRIPTION:
The study design is a three-arm, prospective, pre-post intervention trial. Crohn's Disease (CD) patients at 27-29 weeks of pregnancy will self-select to Arm 1 or Arm 2. Controls will be in Arm 3.

1. Arm 1 (diet-CD): 8-10 weeks of dietary intervention (n=66)
2. Arm 2 (no-diet-CD): usual diet with no diet intervention (n=66)
3. Arm 3 (no-diet-control): unaffected controls at the same gestational stage will follow their usual diet and no intervention (n=66).

The goal of this study is to prospectively test the hypothesis that a non-invasive dietary intervention during the last trimester of pregnancy could beneficially shift the microbiome of CD patients and their babies, hereby promoting a healthier immune system during a critical time of the immune system development. Particularly, the study team will test whether favorable diet-driven changes in the microbiome can lead to a reduced risk of postpartum relapse and lower gut inflammation in the offspring.

Stool, saliva, breast milk and umbilical cord blood samples will be collected, and questionnaires administered. Self-selected participants to Arm 1 will adopt a specified diet, which will be adapted to address specific needs of third trimester pregnancy without compromising the diet principles. Subjects will receive nutritional counseling and training, and compliance to dietary recommendations will be recorded.

Analysis will be performed to correlate dietary change and assessed changes in quality of life with microbial composition in the gut and with circulating markers of inflammation in moms. The study team will also compare the effect of diet vs. non-diet on babies' microbiome and the impact of the early life microbiome in levels of inflammatory markers after 1-year of partum.

This study will help better understand the origin of the initial bacterial colonization in high-risk babies, providing potential intervention targets for primary CD prevention. The study team will also generate an extensive collection of serial samples and longitudinal clinical data, including identification of specific dietary components correlated with certain functional and quantitative bacterial patterns for future investigations. This study will help create new opportunities to foster a healthy microbiome in high risk babies of microbiome and immunity-mediated diseases, thereby hopefully reducing their risk later in life.

ELIGIBILITY:
Inclusion Criteria:

* Capacity to sign informed consent
* At least 18 years old
* Singleton pregnancy of less than 27-29 weeks gestation
* English-speaking

Exclusion Criteria:

* Inability to provide informed consent
* HIV/AIDS
* Multi-fetus pregnancy
* Fetal chromosomal or structural abnormalities
* Active infection (including chorioamnionitis or sepsis)
* Alcohol use disorder
* Diagnosis of diabetes, renal disease, or intrauterine growth restriction
* Non-English speaking
* Active perianal or extraintestinal disease
* Antibiotic or steroid treatment at recruitment
* Scheduled cesarean section prior to gestational week 37

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Change in overall number of proteobacteria | Baseline and 4 Years
  Change in overall number of proteobacteria in pregnant CD patients at 4 years as compared to baseline

SECONDARY OUTCOMES:
Calprotectin level | 4 Years
  Calprotectin is a stool marker of inflammation
Harvey Bradshaw index (HBI) | 4 Years
  Assessments of CD symptom severity
SF-12 | 4 Years
  Quality of life will be assessed using the SF-12.
  Mental and physical functioning is assessed by the Medical Outcomes Study Short Form 12 (SF-12) Health Survey. The questions in the SF-12 target eight dimensions of health and are weighted and summed to provide two composite measures, the Physical Composite Scale and Mental Composite Scale (PCS and MCS). The PCS and MCS are scored to range from 0 to 100, with 0 indicating the lowest level of health and 100 indicating the highest level of health.
The Rome IV Criteria | 3 months
  The Rome IV Criteria for Functional Gastrointestinal Disorders in Infants will be used to assess infant's functional gastrointestinal disorders at 3 months of age. The Rome IV is a validated diagnostic criteria used to improve clinical care in infants and toddlers, adequately diagnose functional gastrointestinal disorders in order to provide proper treatment, and improve homogeneity in research study design.
The Center for Epidemiologic Studies Depression Scale-Revised (CESD-R) | 4 Years
  The CES-D is a 20-item measure assessing symptoms of depression based on a 4-point Likert scale ranging from 0 -3, with higher score indicating more depression.
  and depressive disorder. The symptoms it measures are those defined by the American Psychiatric Association Diagnostic and Statistical Manual (DSM-V) for a major depressive episode.
The Bristol Stool Form Scale | 4 Years
  A validated 7 point scale used extensively in clinical practice and research for classification of stool form. The scale is from 1-7 and a higher score indicates looser stool. A score of 1 is classified as "separate hard lumps, like nuts (hard to pass), while a score of 7 is classified as "Watery, no solid pieces (entirely liquid)."
Alternative Healthy Eating Index | 4 Years
  Alternative Healthy Eating Index (AHEI) - total score ranging from 2.5 (least desirable) to 87.5 (most desirable) dietary pattern

CONTACTS AND LOCATIONS:
Overall Officials: Inga Peter, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Barbara Olendzki, RD,MPH, LDN, Principal Investigator — University of Massachusetts, Worcester; Ana Maldonado-Contreras, PhD, Principal Investigator — University of Massachusetts, Worcester
Locations (2):
- United States (2):
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Icahn School of Medicine at Mount Sinai, New York, New York

IPD SHARING:
Plan to Share IPD: No